CLINICAL TRIAL: NCT04487613
Title: Effect of Moringa Oleifera Capsule in Increasing Breast Milk Volume in Early Postpartum Patients: A Double Blind Randomized Controlled Trial
Brief Title: Effect of Moringa Oleifera Capsule in Increasing Breast Milk Volume in Early Postpartum Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Prof. Vorapong Phupong, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 704/2020
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Postpartum Women

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa oleifera leaf (Active Comparator): Participants received Moringa oleifera leaf 450 mg capsule orally twice daily for 3 days.
  Interventions: Drug: Moringa oleifera leaf
- Placebo (Placebo Comparator): Participants received placebo capsule orally twice daily for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moringa oleifera leaf — 450 mg capsule
  Arms: Moringa oleifera leaf
Drug: Placebo — placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of Moringa oleifera leaf capsule in increasing breast milk volume

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women

Exclusion Criteria:

* Postpartum women with contraindication for breast feeding such as HIV, untreated tuberculosis, on chemotherapeutic drugs, on radioactive drugs, substance abuse.
* Postpartum women with unstable conditions such as postpartum hemorrhage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 88 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Breast milk volume at postpartum day 3 | day 3
  Breast milk volume measuring by weighting the infant fully clothed before and after each feeding with an electronic weigh scale for the period of 24 hours (at postpartum day 3). The sum of weight difference in gram was then converted to breast milk volume in milliliter (1 g = 1 mL).

SECONDARY OUTCOMES:
percentage of good satisfaction | 3 days
  satisfaction evaluated by 5 scales
quality of life scores | 3 days
  Quality of life measuring by Thai version of WHO-QOL questionaire
side effects | 3 days
  percentage of side effects such as headache, nausea/vomiting
Compliance | 3 days
  percentage of complete drug use

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awaliyah SN, Rachmawati IN, Rahmah H. Breastfeeding self-efficacy as a dominant factor affecting maternal breastfeeding satisfaction. BMC Nurs. 2019 Aug 16;18(Suppl 1):30. doi: 10.1186/s12912-019-0359-6. eCollection 2019. PMID 31427892
- [Background] Maharlouei N MD, Pourhaghighi A Medical student, Raeisi Shahraki H PhD, Zohoori D MD, Lankarani KB MD. Factors Affecting Exclusive Breastfeeding, Using Adaptive LASSO Regression. Int J Community Based Nurs Midwifery. 2018 Jul;6(3):260-271. PMID 30035142
- [Background] Frawley J, Adams J, Steel A, Broom A, Gallois C, Sibbritt D. Women's Use and Self-Prescription of Herbal Medicine during Pregnancy: An Examination of 1,835 Pregnant Women. Womens Health Issues. 2015 Jul-Aug;25(4):396-402. doi: 10.1016/j.whi.2015.03.001. Epub 2015 Apr 29. PMID 25935822
- [Background] Zapantis A, Steinberg JG, Schilit L. Use of herbals as galactagogues. J Pharm Pract. 2012 Apr;25(2):222-31. doi: 10.1177/0897190011431636. PMID 22392841
- [Background] Raguindin PF, Dans LF, King JF. Moringa oleifera as a Galactagogue. Breastfeed Med. 2014 Jul-Aug;9(6):323-4. doi: 10.1089/bfm.2014.0002. Epub 2014 Jun 3. No abstract available. PMID 24892837
- [Background] Stohs SJ, Hartman MJ. Review of the Safety and Efficacy of Moringa oleifera. Phytother Res. 2015 Jun;29(6):796-804. doi: 10.1002/ptr.5325. Epub 2015 Mar 24. PMID 25808883
- [Background] Butte NF, Wong WW, Patterson BW, Garza C, Klein PD. Human-milk intake measured by administration of deuterium oxide to the mother: a comparison with the test-weighing technique. Am J Clin Nutr. 1988 May;47(5):815-21. doi: 10.1093/ajcn/47.5.815. PMID 2834941
- [Result] Paritakul P, Ruangrongmorakot K, Laosooksathit W, Suksamarnwong M, Puapornpong P. The Effect of Ginger on Breast Milk Volume in the Early Postpartum Period: A Randomized, Double-Blind Controlled Trial. Breastfeed Med. 2016 Sep;11:361-5. doi: 10.1089/bfm.2016.0073. Epub 2016 Aug 9. PMID 27505611
- [Derived] Fungtammasan S, Phupong V. The effect of Moringa oleifera capsule in increasing breastmilk volume in early postpartum patients: A double-blind, randomized controlled trial. PLoS One. 2021 Apr 6;16(4):e0248950. doi: 10.1371/journal.pone.0248950. eCollection 2021. PMID 33822798